CLINICAL TRIAL: NCT02193204
Title: Chronic Alcohol, Stress Inflammatory Response and Relapse Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1111009349; 1R01AA02009501A (Other: Other Federal Funding)
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Dependence; Depressive Symptomatology
Keywords: Alcohol dependence; Stress; Cytokines; Depressive Symptomatology
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Social Drinkers Depressive Symptoms (Experimental): 30 non-dependent light socially drinking (SD) smokers with depressive symptoms will be recruited to participate in two laboratory sessions (Stress and Neutral / Relaxing). This arm will be exposed to both the personal stress imagery and neutral imagery interventions.
  Interventions: Behavioral: Personal Stress Imagery; Behavioral: Neutral Imagery
- Social Drinkers No Depressive Symptoms (Experimental): 30 non-dependent light socially drinking (SD) smokers without depressive symptoms will be recruited to participate in two laboratory sessions (Stress and Neutral / Relaxing). This arm will be exposed to both the personal stress imagery and neutral imagery interventions.
  Interventions: Behavioral: Personal Stress Imagery; Behavioral: Neutral Imagery
- Alcohol Dependent, Non-Depressive (Experimental): 30 treatment-engaged 28-day abstinent, alcohol dependent (AD) smokers, without Depressive symptoms. All AD subjects will either be admitted to the Clinical Neuroscience Research Unit (CNRU) of the Connecticut Mental Health Center for five weeks of inpatient stay and study participation (inpatient), or they will be scheduled for a two night stay on the CNRU following 3 weeks of abstinence (outpatient). This arm will be exposed to both the personal stress imagery and neutral imagery interventions.
  Interventions: Behavioral: Personal Stress Imagery; Behavioral: Neutral Imagery
- Alchohol Dependent Depressive Symptoms (Experimental): 30 treatment-engaged 28-day abstinent, alcohol dependent smokers with depressive symptoms. All AD subjects will either be admitted to the Clinical Neuroscience Research Unit (CNRU) of the Connecticut Mental Health Center for five weeks of inpatient stay and study participation (inpatient), or they will be scheduled for a two night stay on the CNRU following 3 weeks of abstinence (outpatient). This arm will be exposed to both the personal stress imagery and neutral imagery interventions.
  Interventions: Behavioral: Personal Stress Imagery; Behavioral: Neutral Imagery

INTERVENTIONS:
Behavioral: Personal Stress Imagery — The stress imagery script will be based on participants' description of a recent personal event experienced as "most stressful", and determined as such by rating it above 8 on a 10-point stress scale. These may include breakup with a significant other or job-related stress. A 5-minute 'script' of each scenario will be written using Scene Construction Questionnaires where physiological, bodily sensations regarding the event will be obtained. Scripts will then be recorded onto audiotape for guided imagery in the laboratory sessions.
Behavioral: Neutral Imagery — The neutral script will be developed from a personal non-alcohol-related relaxing situation. A 5-minute 'script' of each scenario will be written using Scene Construction Questionnaires where physiological, bodily sensations regarding the event will be obtained. Scripts will then be recorded onto audiotape for guided imagery in the laboratory sessions.

SUMMARY:
The purpose of this study is to examine potential stress and immune systems adaptations underlying craving and relapse vulnerability in alcohol dependent (AD) individuals and social drinkers (SDs) with and without high levels of depressive symptomatology (+dep / - dep). Using the investigators experimentally validated guided imagery procedure, the investigators propose to examine the response of brain stress and immune systems to personalized guided stressful imagery using subjective, physiological and neurobiological assessments in 60 healthy controls and 60 alcoholic dependent individuals with and without depressive symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* ADs: Male and females, aged 18-50 years, meeting current DSM-IV criteria for alcohol dependence consuming more than 25 drinks / week.
* SDs: Male and females, aged 18-50 years. Must not meet either current or lifetime DSM-IV criteria for alcohol/drug abuse. They must have demonstrated weekly alcohol use over the past year but no more than 25 drinks / month with no occasion of binge drinking (5 or more drinks-men; 4 or more -women).
* ADs and SDs must self-report depression ratings at levels to match one of the two following groups: a) a score of 20 or above in the Center for Epidemiologic Studies - Depression Scale (CES-D), or b) a score between 3 -20 on the CES-D
* Weekly alcohol use as documented by positive urine toxicology screens (AD only).
* Good health as verified by screening examinations and medical and screening
* Able to read English and complete study evaluations.
* All participants must voluntarily provide informed consent and sign the informed consent document.

Exclusion Criteria:

* Meeting current criteria for dependence on another psychoactive substance, excluding nicotine.
* Having any current Axis I psychiatric disorders and requiring treatment/medication for these conditions.
* Having significant underlying medical conditions requiring medication.
* Women who are pregnant or nursing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
cytokine levels | Day 1 and 2, (-25, -5, +5, +15, +30, +45)
  At each of the six time-points (-25, -5, +5, +15, +30, +45), serum cytokine concentrations of IL-6, TNFa, TNFR1, IL-10, IL1-ra, IL-4, IL1beta, and IL-12 will be collected. Levels will be determined by enzyme-linked immuno-sorbent assays using the DuoSet ELISA Development Kit from R&D systems (Minneapolis, MN, USA). Plasma Cortisol and ACTH levels will also be colected and assays will be measured using standard radioimmunoassay procedures.

SECONDARY OUTCOMES:
Alcohol Craving | Day 14, Day 30 and Day 90
  Participants will rate their desire to have an alcoholic drink as well as how anxious they feel at that moment using a10-point visual analog scale (VAS).
Anxiety and Negative Mood | Day 14, Day 30 and Day 90
  Differential Emotion Scale - DES (Izard, 1972): Subjects are required to rate on a 5-point scale the extent to which an emotional word (item) describes the way s/he feels at the current time. Data is collapsed into subscales: anger, anxiety, fear, sadness, joy, and relaxed state.
Alcohol Relapse | 14, 30 and 90 day follow-ups
  Relapse will be defined as a dichotomous variable and any alcohol use during the ninety days post discharge will be coded as relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Fox, PhD, Principal Investigator — Yale University
Locations (1):
- CT Mental Health Center, New Haven, Connecticut, United States